CLINICAL TRIAL: NCT00800462
Title: Comparative Study of the Efficacy and Safety of Muscarinic M3 Receptors Antagonists in the Treatment of Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Magdy Hassouna, MD PhD FRCSC FACS, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-SCI-M3-488
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Spinal Cord Injury; Neurogenic Detrusor Overactivity
MeSH Terms: conditions — Spinal Cord Injuries | interventions — darifenacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxybutynin Cl (Active Comparator)
  Interventions: Drug: Oxybutynin Cl
- Trospium Cl (Active Comparator)
  Interventions: Drug: Trospium Cl
- Darifenacin Hydrogren Bromide (HBr) (Active Comparator)
  Interventions: Drug: Darifenacin Hydrogen Bromide (HBr)

INTERVENTIONS:
Drug: Oxybutynin Cl — 15 mg qd for 3 months
  Other Names: Uromax
  Arms: Oxybutynin Cl
Drug: Trospium Cl — 20mg bid for 3 months
  Other Names: Trosec
  Arms: Trospium Cl
Drug: Darifenacin Hydrogen Bromide (HBr) — 15 mg qd for 3 months
  Other Names: Enablex
  Arms: Darifenacin Hydrogren Bromide (HBr)

SUMMARY:
This is a phase IV, double-blind, multicenter, randomized trial evaluating the efficacy and safety of two M3 receptors antagonists (Trospium Chloride and Darifenacin Hydrobromide) with one standard drug (Oxybutynin Chloride) for treatment of overactive bladder in individuals with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, between 18 and 75 years of age. Female patients of childbearing potential* must have a negative urine pregnancy test result on the day of Screening Visit and practice a reliable method of contraception**

   *A female is considered of childbearing potential unless she is:
   * Postmenopausal for at least 12 months prior to study drug administration;
   * Without a uterus and/or both ovaries; or
   * Has been surgically sterilized for at least 6 months prior to study drug administration.

     **Reliable methods of contraception include:
   * Hormonal methods or intrauterine device in use at least 30 days prior to study drug administration;
   * Barrier methods plus spermicidal in use at least 14 days prior to study drug administration; or
   * Sexual abstinence as a lifestyle.
2. Patients with a neurogenic bladder and detrusor overactivity secondary to a spinal cord injury.

   * Patients with urinary incontinence (minimum of one occurrence per day) despite current treatment. [NOTE: Bladder emptying may be accomplished with straining, intermittent catheterization (IC), spontaneous micturition or leakage episodes.]
3. Patients with serum creatinine within normal limits and normal renal function
4. Patients on a stable dose (minimum one month) of concomitant medication for Neurogenic detrusor overactivity
5. Patients must have adequate cognitive function to understand the requirements of the study, including completing questionnaires and signing a written Informed Consent.

Exclusion Criteria:

1. Female patients who are pregnant (positive urine pregnancy test), planning to become pregnant during the study period, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
2. Patients with a history of transurethral sphincterotomy, bladder neck or prostatic resection, previous bladder surgery including myomectomy or augmentation cystoplasty.
3. Patients with chronic indwelling catheters.
4. Patients with, in the opinion of the Investigator, unstable or stable multiple sclerosis.
5. Patients with known, uncontrolled systemic disease.
6. Patients with evidence of recent alcohol/drug abuse.
7. Patients with urinary retention, gastrointestinal obstructive disorders or uncontrolled narrow-angle glaucoma.
8. Patients with contraindications to Trosec™, Enablex™ and Uromax®.
9. Patients who, in the opinion of the Investigator, have a significant condition or situation that may put the patient at significant risk, confound the study results, or interfere significantly with the patient's participation in the study.
10. Patients with a history of poor cooperation, non-compliance, or unreliability.
11. Patients currently participating in an investigational drug study or who have participated in an investigational drug study within 30 days of the Screening Visit.
12. Patients administered anticholinergics and/or antispasmodic drugs during the course of the study.
13. Patient with hepatic insufficiency.
14. Patient has been administered intravesical botulinum toxin within 6 months prior to the Screening Visit and/or is expected to receive intravesical botulinum toxin during the course of the study.
15. Patient has any medical condition that would interfere with the interpretation of the study results or the conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Incontinence Episodes | 3 days
Adverse Event Reporting | Each Study Visit and Follow-up Phone Call

SECONDARY OUTCOMES:
Urodynamic Study | Baseline and 3 months
Questionnaires | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Hassouna, MD, Principal Investigator — Toronto Rehabilitation Institute
Locations (2):
- Canada (2):
  - University of Manitoba, Health Sciences Centre, Winnipeg, Manitoba
  - Toronto Rehabilitation Institute, Lyndhurst Centre, Toronto, Ontario

REFERENCES:
- See also: Ontario Neurotrauma Foundation — http://www.onf.org